CLINICAL TRIAL: NCT03735680
Title: A Phase 2a, Single-dose, Open-label Study to Evaluate Diagnostic Performance, Safety & Timing of Postdose Imaging of ONM-100, an Intraoperative Fluorescence Imaging Agent for the Detection of Cancer, in Patients With Solid Tumors Undergoing Routine Surgery
Brief Title: A Study to Evaluate ONM-100, an Intraoperative Fluorescence Imaging Agent for the Detection of Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OncoNano Medicine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ON-1002
Record Dates: First submitted 2018-10-24; First posted 2018-11-08 (Actual); Results first posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer; Head and Neck Squamous Cell Carcinoma; Colorectal Cancer; Prostate Cancer; Ovarian Cancer; Urothelial Carcinoma; Non-small Cell Lung Cancer
MeSH Terms: conditions — Breast Neoplasms; Squamous Cell Carcinoma of Head and Neck; Colorectal Neoplasms; Prostatic Neoplasms; Ovarian Neoplasms; Carcinoma, Transitional Cell; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients receiving ONM-100 (Experimental): All patients in this arm will receive ONM-100 for injection and undergo intraoperative imaging.
  Interventions: Drug: ONM-100

INTERVENTIONS:
Drug: ONM-100 — A polymer micelle covalently conjugated to indocyanine green.

SUMMARY:
This study is to evaluate diagnostic performance, safety and timing of post-dose imaging of ONM-100, an intraoperative fluorescence imaging agent for the detection of cancer in patients with solid tumors undergoing routine surgery.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-confirmed diagnosis of primary or recurrent respective tumor type and scheduled to undergo surgical resection
* Part 1: Biopsy-confirmed diagnosis of head and neck squamous cell carcinoma (HNSCC) or breast cancer
* Part 2: Biopsy-confirmed diagnosis of HNSCC, breast cancer, colorectal cancer, prostate cancer, ovarian cancer, urothelial carcinoma and non-small cell lung cancer.
* Part 3: Stage 2 to 4 HNSCC Including T0 or Tx unknown Primary cancers

Exclusion Criteria:

* Histologically diagnosed by an excisional biopsy procedure
* Tumors at sites of which the surgeon would assess that in vivo intraoperative imaging would not be feasible
* Life expectancy <12 weeks
* Hepatic impairment (Child-Pugh score >5) or significant liver disease including active hepatitis or cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trials@OncoNanoMed.com, Study Director — OncoNano Medicine, Inc.
Locations (3):
- United States (3):
  - The University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas - M.D. Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1, Cohort A: Patients were administered a single dose of pegsitacianine (ONM-100) at 1 mg/kg and underwent surgery and fluorescence imaging at 3 ±2 hours post dose.
- Part 1, Cohort B: Patients were administered a single dose of pegsitacianine (ONM-100) at 3 mg/kg for safety evaluation and surgery and imaging at 3 ±2 hours post dose.
- Part 1, Cohort E: Patients were administered a single dose of pegsitacianine (ONM-100) 2 mg/kg and evaluated whether alternate imaging schedules post dose (ie, other than 3 ±2 hours post dose) provided acceptable imaging results at doses ≤3 mg/kg.
- Part 2, Group 2: Patients were administered a single dose of pegsitacianine (ONM-100) at 3 mg/kg. Surgery/imaging time hours to be determined (TBD).
- Part 2, Group 3: Patients were administered a single dose of pegsitacianine (ONM-100) at 1.0 mg/kg. Surgery/imaging time, hours 16-80.
- Part 3: Patients received a single dose of pegsitacianine (ONM-100) at 1 mg/kg administered at 24 ±8 hours prior to surgery.
Period: Overall Study
Arm/Group | Part 1, Cohort A | Part 1, Cohort B | Part 1, Cohort E | Part 2, Group 2 | Part 2, Group 3 | Part 3
Started | 3 | 3 | 3 | 4 | 6 | 11
Completed | 3 | 2 | 2 | 4 | 6 | 10
Not Completed | 0 | 1 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Patient unable or unwilling to continue | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1, Cohort A: Patients were administered a single dose of pegsitacianine (ONM-100) at 1.0 mg/kg and underwent surgery and fluorescence imaging at 3 ±2 hours post dose.
- Part 1, Cohort B: Patients were administered a single dose of pegsitacianine (ONM-100) at 3.0 mg/kg and underwent surgery and fluorescence imaging at 3 ±2 hours post dose.
- Part 1, Cohort E: Patients were administered a single dose of pegsitacianine (ONM-100) at 2 mg/kg and underwent surgery and fluorescence imaging at 6 ±3 hours post dose.
- Part 2, Group 2: Patients were administered a single dose of pegsitacianine (ONM-100) at 3 mg/kg and underwent surgery and fluorescence imaging at a time to be determined post dose.
- Part 2, Group 3: Patients were administered a single dose of pegsitacianine (ONM-100) at 1 mg/kg and underwent surgery and fluorescence imaging at 16-80 hours post dose.
- Part 3: Patients were administered a single dose of pegsitacianine (ONM-100) at 1 mg/kg and underwent surgery and fluorescence imaging at 24 ±8 hours post dose.
- Total: Total of all reporting groups
Arm/Group | Part 1, Cohort A | Part 1, Cohort B | Part 1, Cohort E | Part 2, Group 2 | Part 2, Group 3 | Part 3 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 6 | 11 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (8.19) | 63.7 (3.79) | 59.3 (15.31) | 65.5 (5.07) | 59.8 (4.71) | 59.8 (10.26) | 60.5 (8.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 1 | 0 | 3 | 8
  Male | 1 | 2 | 2 | 3 | 6 | 8 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 1 | 0 | 3
  Not Hispanic or Latino | 1 | 2 | 3 | 4 | 5 | 10 | 25
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 0 | 1 | 2 | 5
  White | 3 | 3 | 1 | 3 | 5 | 7 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 4 | 6 | 11 | 30
Patients receiving pegsitacianine (ONM-100) [Count of Participants; unit: Participants] | 3 | 3 | 3 | 4 | 6 | 11 | 30

OUTCOME MEASURES:

1. Primary Outcome: Measure Mean Fluorescence Intensity of Histologically Confirmed Tumor vs Normal Tissue in Patients Undergoing Routine Surgery [Tumor to Background Ratio (TBR)]
Description: Part 1: Evaluate the dose(s) at which ONM-100 fluorescence imaging is feasible at 3±2 hours post dose.
  Part 2: Verify the safety and diagnostic performance of ONM-100 compared to standard pathology at the dose(s) and imaging schedule(s) post dose selected from Part 1 for the detection of primary tumors and the metastatic lymph nodes in a variety of solid cancers (which could have included HNSCC, breast cancer, colorectal cancer, urothelial cancer, prostate cancer, ovarian cancer, and/or non-small cell lung carcinoma [NSCLC]).
  Part 3: Assess the safety and efficacy (sensitivity and positive predictive value [PPV] of ONM-100 for intraoperative imaging during HNSCC surgery.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Part 1, Cohort A: All patients in this arm received a single IV administration of ONM-100) at 1 mg/kg.
- Part 1, Cohort B; Part 2, Group 2: All patients in this arm received a single IV administration of ONM-100 at 3 mg/kg.
- Part 1, Cohort E: All patients in this arm received a single IV administration of ONM-100 at 2 mg/kg.
- Part 2, Group 3; Part 3: All patients in this arm received a single IV administration of ONM-100 at 1 mg/kg.
Arm/Group | Part 1, Cohort A | Part 1, Cohort B | Part 1, Cohort E | Part 2, Group 2 | Part 2, Group 3 | Part 3
Number analyzed (Participants) | 1 | 3 | 3 | 4 | 6 | 11
ratio | 1.098 (0) | 4.022 (2.8139) | 2.280 (1.6393) | 4.110 (1.2527) | 3.007 (1.3822) | 2.608 (2.5936)

2. Primary Outcome: Incidence Rate of All Treatment-emergent Adverse Events (TEAEs) From Time of ONM-100 Administration Through Day 28
Description: Evaluate safety at the dose(s) used to assess imaging feasibility and select the dose(s) and imaging schedule(s) post dose that are safe and provide optimal imaging of solid tumors and metastatic lymph nodes; the dose and time post dose chosen for the detection of primary tumors and metastatic lymph nodes could be the same or different.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Groups:
- Part 1, Cohort A; Part 2, Group 3; Part 3: Patients were administered a single IV infusion of ONM-100 at a dose of 1 mg/kg.
- Part 1, Cohort B: Patients were administered a single IV infusion of OMN-100 at a dose of 3 mg/kg.
- Part 1, Cohort E: Patients were administered a single IV infusion of OMN-100 at a dose of 2 mg/kg.
- Part 2, Group 2: Patients were administered a single IV infusion of ONM-100 at a dose of 3 mg/kg.
Arm/Group | Part 1, Cohort A | Part 1, Cohort B | Part 1, Cohort E | Part 2, Group 2 | Part 2, Group 3 | Part 3
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 6 | 11
Participants | 2 | 3 | 2 | 4 | 6 | 9

3. Secondary Outcome: Evaluate Pharmacokinetic Parameters: Cmax
Description: Evaluate the maximum plasma concentration (Cmax) of ONM-100 at the dose(s) and imaging schedule(s) post dose used to assess optimal imaging at doses of 1 mg/kg, 2 mg/kg and 3 mg/kg.
Time Frame: 6 days
Population: The PK analysis population is comprised 19 patients for whom concentration data were available. Due to sparse plasma concentrations for the majority of patients, with the exception of Cmax and Tmax, it was not possible to estimate all parameters for all patients.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Groups:
- Patients Receiving ONM-100 a Dose of 1 mg/kg: All patients in the study who received a single IV administration of ONM-100 at 1 mg/kg.
- Patients Receiving ONM-100 at a Dose of 2 mg/kg: All patients in the study who received a single IV administration of ONM-100 at 2 mg/kg.
- Patients Receiving ONM-100 at a Dose of 3 mg/kg: All patients in the study who received a single IV administration of ONM-100 at 3 mg/kg.
Arm/Group | Patients Receiving ONM-100 a Dose of 1 mg/kg | Patients Receiving ONM-100 at a Dose of 2 mg/kg | Patients Receiving ONM-100 at a Dose of 3 mg/kg
Number analyzed (Participants) | 9 | 3 | 6
μg/mL | 26.5 (16.0) | 52.2 (13.0) | 79.5 (30.0)

4. Secondary Outcome: Evaluate Pharmacokinetic Parameters: Tmax
Description: Evaluate the time to Cmax (Tmax) of ONM-100 at the dose(s) and imaging schedule(s) post dose used to assess optimal imaging in Part 1 and Part 2.
Time Frame: 6 days
Population: The PK analysis population comprised 19 patients for whom concentration data were available. Due to sparse plasma concentrations for the majority of patients, with the exception of Cmax and Tmax, it was not possible to estimate all parameters for all patients.
Measure: Median (Full Range); unit: hr
Groups:
- ONM-100 at Dose of 1 mg/kg: All patients in this arm received IV administration of ONM-100 at a dose of 1 mg/kg.
- ONM-100 at a Dose of 2 mg/kg: All patients in this arm received IV administration of ONM-100 at a dose of 2 mg/kg.
- ONM-100 at a Dose of 3 mg/kg: All patients in this arm received IV administration of ONM-100 at a dose of 3 mg/kg.
Arm/Group | ONM-100 at Dose of 1 mg/kg | ONM-100 at a Dose of 2 mg/kg | ONM-100 at a Dose of 3 mg/kg
Number analyzed (Participants) | 9 | 3 | 6
hr | 0.25 [0.22 to 1.12] | 0.31 [0.27 to 7.35] | 0.31 [0.23 to 0.37]

5. Secondary Outcome: Evaluate Pharmacokinetic Parameters: AUC
Description: Evaluate the Area under the time-concentration curve [AUC] of ONM-100 at 1 mg/kg, 2 mg/kg, and 3 mg/kg doses.
Time Frame: 6 days
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr x μg/mL
Groups:
- ONM-100 at a Dose of 1 mg/kg: Patients receiving a single IV administration of ONM-100 at 1 mg/kg.
- ONM-100 at a Dose of 2 mg/kg: Patients received a single IV administration of ONM-100 at 2 mg/kg.
- ONM-100 at a Dose of 3 mg/kg: Patients receiving a single IV administration of ONM-100 at 3 mg/kg.
Arm/Group | ONM-100 at a Dose of 1 mg/kg | ONM-100 at a Dose of 2 mg/kg | ONM-100 at a Dose of 3 mg/kg
Number analyzed (Participants) | 9 | 3 | 6
hr x μg/mL | 433 (127) | 1509 (80.1) | 2067 (38.4)

6. Secondary Outcome: Evaluate Pharmacokinetic Parameters: CL
Description: Evaluate Total body clearance [CL] of ONM-100 at the dose(s) and imaging schedule(s) post dose used to assess optimal imaging in Part 1 and Part 2.
Time Frame: 6 days
Population: The PK analysis population comprised 19 patients for whom concentration data were available. Due to the sparse plasma concentrations for the majority of patients, with the exception of Cmax and Tmax, it was not possible to estimate all parameters for all patients.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | ONM-100 at a Dose of 1 mg/kg | ONM-100 at a Dose of 2 mg/kg | ONM-100 at a Dose of 3 mg/kg
Number analyzed (Participants) | 2 | 0 | 2
L/hr | 0.053 (2.57) |  | 0.053 (70.5)

7. Secondary Outcome: Evaluate Pharmacokinetic Parameters: Vz
Description: Evaluate the Volume of distribution [Vz] of ONM-100 at the dose(s) and imaging schedule(s) post dose used to assess optimal imaging in Part 1 and Part 2.
Time Frame: 6 days
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | ONM-100 at Dose of 1 mg/kg | ONM-100 at a Dose of 2 mg/kg | ONM-100 at a Dose of 3 mg/kg
Number analyzed (Participants) | 2 | 0 | 2
L | 3.78 (33.9) |  | 5.32 (82.9)

8. Secondary Outcome: Evaluate Pharmacokinetic Parameters: t1/2
Description: Evaluate the Terminal elimination half-life [t1/2] of ONM-100 at the dose(s) and imaging schedule(s) post dose used to assess optimal imaging in Part 1 and Part 2.
Time Frame: 6 days
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | ONM-100 at Dose of 1 mg/kg | ONM-100 at a Dose of 2 mg/kg | ONM-100 at a Dose of 3 mg/kg
Number analyzed (Participants) | 2 | 0 | 2
hr | 49.0 (36.7) |  | 69.4 (8.80)

ADVERSE EVENTS:
Time Frame: The total collection period for each subject was approximately one month.
Groups:
- Part 1, Cohort A; Part 2, Group 3; Part 3: ONM-100 at dose of 1 mg/kg.
- Part 1, Cohort B; Part 2, Group 2: ONM-100 at dose of 3 mg/kg.
- Part 1, Cohort E: ONM-100 at dose of 2 mg/kg.
Arm/Group | Part 1, Cohort A | Part 1, Cohort B | Part 1, Cohort E | Part 2, Group 2 | Part 2, Group 3 | Part 3
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/4 | 0/6 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/3 | 0/3 | 1/4 | 0/6 | 3/11
Other Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 2/3 | 4/4 | 4/6 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1, Cohort A (N=3) | Part 1, Cohort B (N=3) | Part 1, Cohort E (N=3) | Part 2, Group 2 (N=4) | Part 2, Group 3 (N=6) | Part 3 (N=11)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1, Cohort A (N=3) | Part 1, Cohort B (N=3) | Part 1, Cohort E (N=3) | Part 2, Group 2 (N=4) | Part 2, Group 3 (N=6) | Part 3 (N=11)
Infusion-related reaction (Injury, poisoning and procedural complications) | 1 (2) | 2 (4) | 0 (0) | 3 (6) | 4 (8) | 7 (24)
Buttock injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dizziness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensory disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/80/NCT03735680/Prot_000.pdf